CLINICAL TRIAL: NCT03076567
Title: Discovery and Validation of Plasma DNA Methylation Biomarker for Detection of Stomach Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917063; 17-C-N063
Record Dates: First submitted 2017-03-09; First posted 2017-03-10 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Stomach Cancer; Gastric Cancer
Keywords: Epidemiology; Cancer; Methylation; Genetics; Screening
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Testing pre-existing serum samples from 2 ongoing studies covered by other SSIRB approvals - OH95-C-N027-G (Esophageal CA Genetic Studies) and PH99-C-N031-H (Nutritional Intervention Trials in Linxian China - Continued Follow-Up)

GROUPS / COHORTS (2):
- case: Stomach cancer cases from two previously conducted studies in China
- control: Controls from two previously conducted studies in China

SUMMARY:
Background:

Stomach cancer is common around the world. The US is a low-risk region. But the 5-year survival rate in the US is low. This is because the cancer is usually in a late stage by the time it is diagnosed. One way to detect it earlier is to screen many people with a procedure called endoscopy. But this may not be feasible in low-risk or developing countries. Researchers want to find a biomarker for early-stage disease to help them create an effective way of screening. DNA methylation is a chemical modification of DNA. It generates a signal for certain cancers, including stomach cancer. Researchers want to find a blood-based DNA methylation marker for stomach cancer.

Objective:

To study plasma DNA methylation as a potential biomarker for detection of stomach cancer.

Eligibility:

Participants from 2 studies already done in China

Design:

Researchers will use blood samples from participants in the 2 studies. The blood was collected in 1999/2000. They will use samples from some who developed stomach cancer between those years and 2006. The other samples will be from some who stayed cancer free in that time.

Participants already gave written informed consent.

Researchers will take DNA from the samples. They will look for methylation.

DETAILED DESCRIPTION:
Despite markedly declining incidence in recent decades, almost one million new cases of stomach cancer were estimated to have occurred in 2012, making it the fifth most common malignancy in the world after lung, breast, colorectal, and prostate cancer. More than 70% of cases (677,000 cases) occur in developing countries, and half occur in Eastern Asia (mainly in China). Although North America is considered to be a low-risk region, 22,000 cases are diagnosed in the US each year. Five-year survival for 2005-2011 in the US was less than 30%, since stomach cancer is generally asymptomatic in early stages and has often metastasized by the time of diagnosis. In contrast, 5-year survival rates are almost 70% in South Korea and Japan where mass screening programs have been implemented and a large proportion of stomach cancer is detected in early stages. UGI endoscopy has been considered as the gold standard for diagnosis of stomach cancer but endoscopy-based mass screening may not be feasible in relatively low-risk or less developed regions. Therefore, identification of biomarkers for early stage disease is crucial to in the development of effective screening strategies. With the recent advances in cancer genetics and assay technologies, this is an opportune time to discover minimally invasive, specific, and cost-effective biomarkers.

A surprising discovery from the large scale cancer genome projects such as TCGA was the enormous variation in mutational patterns both across and within individual tumor types. Even the most commonly mutated genes were typically altered in less than half of cases of a given cancer. The two most frequently mutated driver genes in stomach cancer, TP53 (tumor protein p53) and ARID1A (AT rich interactive domain 1A), were mutated in only 44% and 17% of cases, respectively. Mutation rates for the remaining stomach cancer driver genes were even lower. Importantly, mutations of these genes are often spread across several exons which complicates detection of DNA-based sequence variation, since large numbers of samples and extensive genotyping will be required to achieve adequate sensitivity and power. In contrast, DNA methylation, which is a chemical modification of CpG dinucleotides that does not alter base pair sequence, generates a more robust signal as compared to genetic alterations. For example, methylation in the Stratifin promoter was found in 96% (24/25) of breast carcinomas, 83% (15/18) of ductal carcinoma in situ, and 38% (3/8) of benign atypical hyperplasias, but was absent in breast tissues from healthy individuals, which suggests that methylation status of this locus is an early event of breast cancer that could serve as a breast cancer biomarker. Aberrant DNA methylation occurs in an early phase of carcinogenesis and contributes to development and progression. Notably, a comprehensive molecular characterization of 295 primary stomach cancers in TCGA classified the tumors into four molecular subtypes. All four types exhibited DNA hypermethylation to various degrees, with one type more heavily methylated than any other tumor group previously analyzed in TCGA. Moreover, other studies have also suggested that aberrant methylation may be associated with various pre-malignant conditions like Helicobacter pylori infection, severe gastritis, intestinal metaplasia, and dysplasia, implying a role for an epigenetic field effect which may reflect the earliest steps in neoplastic transformation of the stomach. Importantly, hypermethylation can be detected in circulating cell-free DNA (cfDNA) which is thought to be derived from preneoplastic or tumor tissues. Efforts to discover blood-based DNA methylation markers are underway in various types of cancers. In particular, plasma methylated SEPT9 DNA has been evaluated for detection of colorectal cancer, and a commercialblood test for this is under review for approval by the US Food and Drug Administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

Data samples already exist from 2 other IRB approved studies (OH99-C-N031, OH95-C-N027)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nutrition Intervention Trials (NIT) - Community Sample Shanxi - Hospital and community samples@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Relation of DNA methylation marakers to gastric cancer status | ongoing
  Relation of markers tested to cancer

CONTACTS AND LOCATIONS:
Overall Officials: Alisa M Goldstein, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States